CLINICAL TRIAL: NCT01488344
Title: A Single-arm, Open Label, Multi-center Phase I/II Trial to Assess the Safety and Efficacy of BIBF 1120 Added to Low-dose Cytarabine in Elderly Patients With AML Unfit for an Intensive Induction Therapy
Brief Title: Phase I/II Trial: BIBF 1120 Added to Low-dose Cytarabine in Elderly Patients With Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM10_0014; 2011-001086-41 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-12-08 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: triple kinase inhibitor BIBF1120

INTERVENTIONS:
Drug: triple kinase inhibitor BIBF1120 — triple kinase inhibitor BIBF1120 is given in addition to low-dose cytarabine

SUMMARY:
RATIONALE: Low-dose cytarabine works in a minority of elderly patients with an acute myeloid leukemia unfit for intensive induction therapy by killing of leukemia cells. Addition of BIBF1120 to low-dose cytarabine might enhance the killing of leukemia cells.

PURPOSE: This phase I / II trial is studying how safe BIBF1120 can be combined with low-dose cytarabine (phase I) and how well the combination of low-dose cytarabine and BIBF1120 works in elderly patients with acute myeloid leukemia unfit for intensive chemotherapy (phase II).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML (except APL) according to the FAB or WHO classification, including AML evolving from MDS or other hematological diseases and AML after previous cytotoxic therapy or radiation (secondary AML), with medical contraindications against or not willing to receive a standard induction and consolidation therapy.
* Bone marrow aspirate or biopsy must contain > 20% blasts of all nucleated cells. In AML FAB M6 ≥ 30% of non-erythroid cells in the bone marrow must be leukemic blasts. In patients with 20-30% blasts, the indication for a treatment with hypomethylating agents (5-azacitidine or decitabine) should be considered prior to inclusion into the trial.
* Age ≥ 60 years
* Informed consent, personally signed and dated to participate in the study
* Male patients enrolled in this trial must use adequate barrier birth control measures during the course of treatment and for at least 3 months after the last administration of study therapy (low-dose cytarabine and/or BIBF 1120).

Exclusion Criteria:

* Patients with 20-30% bone marrow blasts which are qualifying for and consenting into a therapy with hypomethylating agents
* Patients who are eligible for and consenting into a standard chemotherapy
* Known central nervous system manifestation of AML
* Inadequate liver function (ALT and AST ≥ 2.5 x ULN) if not caused by leukemic infiltration
* Known chronically active hepatitis C infection or acute hepatitis
* Chronically impaired renal function (creatinin clearance < 30 ml/min)
* Uncontrolled hypertension with a resting pressure systolic > 160 mmHg or diastolic > 95 mmHg despite adequate treatment
* severe trauma or surgery within 4 weeks of study entry
* severe, non-healing wounds, ulcer or fracture
* Uncontrolled active infection
* Concurrent malignancies other than AML or other severe diseases which in the opinion of the investigator are likely to influence the endpoint assessment
* Hypersensitivity to cytarabine (not including drug fever or exanthema)
* Previous treatment of AML except hydroxyurea up to 24 hours before study medication
* Previous therapy with tyrosine kinase inhibitors or angiogenesis inhibitors
* Parallel participation in another clinical trial for the same indication. Eligibility of patients with investigational drug therapy outside of this trial during or within 4 weeks of study entry should be discussed with the study office prior to study entry
* Any severe concomitant condition, which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Phase I: defining maximum tolerated dose (MTD) | 4 weeks
Phase II: overall response rate (ORR) | up to 6 month

SECONDARY OUTCOMES:
Complete remission (CR) rate | up to 12 month
overall survival (OS) | up to 12 month
relapse-free survival (RFS)of the responding patients | up to 12 month
number of participants with adverse events as a measure of safety and tolerability | up to 12 month
ORR rate of the Flt3-mutated patients versus the Flt3-wildtype patients | up to 12 month
CR rate of the Flt3-mutated patients versus the Flt3-wildtype patients | up to 12 month
OS of the Flt3-mutated patients versus the Flt3-wildtype patients | up to 12 month
time to response (CR, CRp, CRi) of the responding patients | up to 12 month
  CRp = complete remission with incomplete platelet recovery CRi = complete remission with incomplete neutrophil recovery

CONTACTS AND LOCATIONS:
Overall Officials: Utz Krug, MD, Principal Investigator — University Hospital Münster, Medizinische Klinik und Poliklinik A
Locations (1):
- Universitätsklinikum Münster, Medizinische Klinik und Poliklinik A, Münster, Germany

REFERENCES:
- [Derived] Berdel AF, Koch R, Gerss J, Hentrich M, Peceny R, Bartscht T, Steffen B, Bischoff M, Spiekermann K, Angenendt L, Mikesch JH, Kewitz T, Butterfass-Bahloul T, Serve H, Lenz G, Berdel WE, Krug U, Schliemann C. A randomized phase 2 trial of nintedanib and low-dose cytarabine in elderly patients with acute myeloid leukemia ineligible for intensive chemotherapy. Ann Hematol. 2023 Jan;102(1):63-72. doi: 10.1007/s00277-022-05025-0. Epub 2022 Nov 18. PMID 36399194
- [Derived] Schliemann C, Gerss J, Wiebe S, Mikesch JH, Knoblauch N, Sauer T, Angenendt L, Kewitz T, Urban M, Butterfass-Bahloul T, Edemir S, Vehring K, Muller-Tidow C, Berdel WE, Krug U. A Phase I Dose Escalation Study of the Triple Angiokinase Inhibitor Nintedanib Combined with Low-Dose Cytarabine in Elderly Patients with Acute Myeloid Leukemia. PLoS One. 2016 Oct 7;11(10):e0164499. doi: 10.1371/journal.pone.0164499. eCollection 2016. PMID 27716819